CLINICAL TRIAL: NCT01876134
Title: The Diagnostic Role of Cystein-rich Protein 61 (Cyr61) in Acute Kidney Injury: Correlation With the Harmonic Analysis of Arterial Pressure Pulse Waves.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201210055RIC
Record Dates: First submitted 2013-06-10; First posted 2013-06-12 (Estimated); Last update posted 2013-06-12 (Estimated); Status verified 2013-06

CONDITIONS: Consecutive Incident Adult Patients Undergoing Elective Cardiac Surgery
Keywords: Cardiac surgery; Acute kidney injury; Cyr-61; Pulse wave analysis
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Biospecimen Retention: Samples Without DNA — Urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Elective cardiac surgery

SUMMARY:
Acute kidney injury (AKI) is a common heterogeneous disease that complicates several medical and surgical conditions. Recent studies have demonstrated that the occurrence of AKI significantly increase the risk of adverse outcomes. Despite the advanced in modern medicine, the interventions for AKI are not improved. One major reason of the failure to shift therapeutic progress is the clinicians' widespread dependence upon serum creatinine, an unreliable marker during acute changes of renal function, for the diagnosis of AKI.

In the past decade, over 20 unique biomarkers of AKI had been explored. Among them, neutrophil gelatinase-associated lipocalin (NGAL), interleukin-18 (IL-18), and kidney injury molecule-1 (KIM-1) have received the most interest. None of them, however, is an idea one.

Cysteine-rich protein 61 (Cyr61), a secreted matrix-associated heparin-binding protein, belongs to the "CCN" family. It regulates a broad spectrum of cellular activities, including cell adhesion, migration, proliferation, survival, differentiation, apoptosis, angiogenesis, and extracellular matrix production of multiple cell types. By the kidney ischemic/reperfusion injury animal model, Cyr61 gene was found to be rapidly up-regulated in the renal outer medulla. That portion of the kidney is corresponding to the area of marginally oxygenated under normal condition and most tubular injury following renal ischemic/reperfusion injury.18 Elevation of Cyr61 protein was detected in the kidney and also in urine following injury, making it a potential marker of AKI.

Additionally, pulse diagnosis is an integrative part of traditional Chinese medicine. With spectral analysis of the pulse waves, researchers started to observe the pulse wave harmonics. An in vivo study of rats revealed that ligating one or both of the renal arteries significantly reduced the second harmonic component of the pressure pulse at the caudate artery. Ligating the artery toward the spleen prominently reduced the third harmonics component of the pulse. Analysis of the harmonics in the spectrum of the arterial pressure wave revealed that individual organs might have their own natural frequencies. These observations suggested that individual vascular beds exert independent, frequency-specific, effects on the peripheral pressure wave.

Among different etiologies, cardiac surgery is an important cause of AKI. It has been shown that AKI after cardiac surgery is relatively highly prevalent and prognostically important. Cardiac surgery is usually performed with the use of extracorporeal cardiopulmonary bypass machine ('on-pump').

Based on the evidence from cell culture study and animal study in the literature, we hypothesize that Cyr61 is rapidly increased in the urine after AKI. We thus design this project to evaluate study the diagnostic role and clinical application of Cyr61 in AKI. We will conduct a prospective cohort study to evaluate the changes of urinary Cyr61 in patients undergoing cardiac surgery. Cyr61 may serve a good biomarker for the early diagnosis of patients with AKI, either singly or in combination with NGAL. By the way, we also try to correlate the changes in those biomarker with a potential new tool：harmonic analysis of arterial pressure pulse waves. We have special interest in following the time course of changes in biomarker and correlate with changes in pulse analysis. Physiological parameters of vascular compliance and regional blood oxygen saturation will be correlated concurrently. It is hoped that early detection of AKI will lead to earlier intervention, thus enhancing our ability to develop beneficial therapies.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is a common heterogeneous disease that complicates several medical and surgical conditions. Recent studies have demonstrated that the occurrence of AKI significantly increase the risk of adverse outcomes. Despite the advanced in modern medicine, the interventions for AKI are not improved. One major reason of the failure to shift therapeutic progress is the clinicians' widespread dependence upon serum creatinine, an unreliable marker during acute changes of renal function, for the diagnosis of AKI.

In the past decade, over 20 unique biomarkers of AKI had been explored. Among them, neutrophil gelatinase-associated lipocalin (NGAL), interleukin-18 (IL-18), and kidney injury molecule-1 (KIM-1) have received the most interest. None of them, however, is an idea one.

Cysteine-rich protein 61 (Cyr61), a secreted matrix-associated heparin-binding protein, belongs to the "CCN" family. It regulates a broad spectrum of cellular activities, including cell adhesion, migration, proliferation, survival, differentiation, apoptosis, angiogenesis, and extracellular matrix production of multiple cell types. By the kidney ischemic/reperfusion injury animal model, Cyr61 gene was found to be rapidly up-regulated in the renal outer medulla. That portion of the kidney is corresponding to the area of marginally oxygenated under normal condition and most tubular injury following renal ischemic/reperfusion injury.18 Elevation of Cyr61 protein was detected in the kidney and also in urine following injury, making it a potential marker of AKI.

Additionally, pulse diagnosis is an integrative part of traditional Chinese medicine. With spectral analysis of the pulse waves, researchers started to observe the pulse wave harmonics. An in vivo study of rats revealed that ligating one or both of the renal arteries significantly reduced the second harmonic component of the pressure pulse at the caudate artery. Ligating the artery toward the spleen prominently reduced the third harmonics component of the pulse. Analysis of the harmonics in the spectrum of the arterial pressure wave revealed that individual organs might have their own natural frequencies. These observations suggested that individual vascular beds exert independent, frequency-specific, effects on the peripheral pressure wave.

Among different etiologies, cardiac surgery is an important cause of AKI. It has been shown that AKI after cardiac surgery is relatively highly prevalent and prognostically important. Cardiac surgery is usually performed with the use of extracorporeal cardiopulmonary bypass machine ('on-pump').

Based on the evidence from cell culture study and animal study in the literature, we hypothesize that Cyr61 is rapidly increased in the urine after AKI. We thus design this project to evaluate study the diagnostic role and clinical application of Cyr61 in AKI. We will conduct a prospective cohort study to evaluate the changes of urinary Cyr61 in patients undergoing cardiac surgery. Cyr61 may serve a good biomarker for the early diagnosis of patients with AKI, either singly or in combination with NGAL. By the way, we also try to correlate the changes in those biomarker with a potential new tool：harmonic analysis of arterial pressure pulse waves. We have special interest in following the time course of changes in biomarker and correlate with changes in pulse analysis. Physiological parameters of vascular compliance and regional blood oxygen saturation will be correlated concurrently. It is hoped that early detection of AKI will lead to earlier intervention, thus enhancing our ability to develop beneficial therapies.

ELIGIBILITY:
Inclusion Criteria:

All consecutive incident adult patients undergoing elective cardiac surgery (including coronary artery bypass graft, valve surgery, and correction of congenital heart diseases)

Exclusion Criteria:

age younger than 20 years or older than 80 years; pregnant woman; emergent cardiac surgery; use of intra-aortic balloon pump or extracorporeal membrane oxygenation after surgery, pre-existing severe renal insufficiency (defined as estimated glomerular filtration rate 15 cc/min or less by the Modification of Diet in Renal Disease study equation36); patients with end-stage renal disease under maintenance hemodialysis, peritoneal dialysis, or receiving kidney transplantation; use of radiocontrast ≤24 h prior to the surgery; use of nephrotoxic drugs before or during the surgery

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive incident adult patients undergoing elective cardiac surgery (including coronary artery bypass graft, valve surgery, and correction of congenital heart diseases)
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2013-04; Primary Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Acute kidney injury | 1 week after cardiac surgery
  development of AKI within 1 week after cardiac surgery

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Fu Lai, MD, Study Director — Division of Nephrology, Department of Internal medicine, National Taiwan University Hospital